CLINICAL TRIAL: NCT00938301
Title: A Phase 1, Placebo-Controlled, Crossover Study To Evaluate The Safety, Tolerability And Pharmacokinetics Of PF-04455242 After First-Time Administration Of Single Ascending Doses To Healthy Adult Subjects
Brief Title: A First In Human Study To Evaluate The Safety, Tolerability And Pharmacokinetics Of PF-04455242 In Single Rising Doses In Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B1071001
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Bipolar Depression
Keywords: healthy volunteer, first in human, safety and tolerability
MeSH Terms: conditions — Bipolar Disorder | interventions — 2-methyl-N-((2'-(pyrrolidin-1-ylsulfonyl)biphenyl-4-yl)methyl)propan-1-amine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Active Comparator): 2 cohorts will recieve single rising doses of PF-04455242 or placebo in a cross-over fashion.
  Interventions: Drug: PF-04455242
- Placebo (Placebo Comparator): 2 cohorts will receive single rising doses of PF-04455242 or placebo in a cross-over fashion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04455242 — Powder-in Capsule (EP-PIC), will be used to administer doses from 0.5 mg up to and including 56 mg of a single rising dose over 3 treatment periods receiving two doses of PF-04455242 and one dose of placebo. A one-week (minimum) washout will separate each treatment period.
  Arms: Treatment
Drug: Placebo — PIC matching in appearance to PF-04455242 will be used to administer placebo.
  Arms: Placebo

SUMMARY:
The purpose of this first in human (FIH) study is to investigate the safety, tolerability, pharmacokinetics ( how the body handles the drug) and pharmacodynamics (how the drug affects the body) of PF-04455242-01 in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female of non-childbearing potential between the ages of 18 and 55 years.
* Body Mass Index (BMI) of approximately 18 to 30 kg/m2; and a total body weight >50 kg (>110 lbs).
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

* Evidence or history of clinically significant medical condition or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of screening).
* Use of tobacco- or nicotine-containing products within 3 months of screening or a positive urine or blood cotinine at screening.
* A positive urine drug screen. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single doses will include neurological assessment, vital signs and adverse event reporting during inpatient stay. | Daily
Physical exam | Screening, End of Trial (EOT), and Follow Up (F/U)
Clinical safety laboratory results | Screening, Day 0 (D0), D2, F/U
12-lead ECGs | Screening, D1, D2, F/U
Maximum plasma concentration (Cmax), time to reach maximum concentration (Tmax), area under the concentration-time curve (AUC) and terminal half-life (t1/2) . | 0 hr (predose) then 0.5-1 hr for the next 12 hrs postdose on D1, then 24, 36, 48, & 72 hrs postdose

SECONDARY OUTCOMES:
Likert and Drug Effect Questionnaire (DEQ) questionnaires | 0 hr (predose) then 1, 2, 3, 4, 6 ,8, & 12 hrs (postdose) on D1, then 24 hrs (postdose) on D2

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1071001&StudyName=A%20First%20In%20Human%20Study%20To%20Evaluate%20The%20Safety%2C%20Tolerability%20And%20Pharmacokinetics%20Of%20PF-04455242%20In%20Single%20Rising%20Doses%20In%20Healthy%20Ad